CLINICAL TRIAL: NCT07082738
Title: A Multicentre, Parallel-group, Phase IIb, Randomised, Double-blind, Placebo-controlled, 4-Arm, 24-Week Study to Evaluate the Efficacy and Safety of AZD6793 Tablets in Adult Participants With Moderate to Very Severe Chronic Obstructive Pulmonary Disease (PRESTO)
Brief Title: A Study to Investigate the Effect of AZD6793 in Participants With Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Acronym: PRESTO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7860C00006
Record Dates: First submitted 2025-06-11; First posted 2025-07-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Moderate COPD; Severe COPD; Very Severe COPD; chronic obstructive pulmonary disease; AZD6793; IRAK4
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a ratio of 1:1:1:1 to receive Dose 1 of AZD6793, Dose 2 of AZD6793, Dose 3 of AZD6793 or matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose 1 of AZD6793 (Experimental): Approximately 290 participants will be randomized to receive Dose 1 of AZD6793
  Interventions: Drug: AZD6793
- Dose 2 of AZD6793 (Experimental): Approximately 290 participants will be randomized to receive Dose 2 of AZD6793
  Interventions: Drug: AZD6793
- Dose 3 of AZD6793 (Experimental): Approximately 290 participants will be randomized to receive Dose 3 of AZD6793
  Interventions: Drug: AZD6793
- Matching Placebo (Placebo Comparator): Approximately 290 participants will be randomized to receive Matching Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD6793 — Oral dosage
  Arms: Dose 1 of AZD6793; Dose 2 of AZD6793; Dose 3 of AZD6793
Other: Placebo — Oral dosage
  Arms: Matching Placebo

SUMMARY:
This Phase IIb dose-ranging study will evaluate the efficacy and safety of 3 different doses of AZD6793 compared with placebo tablets in participants with moderate to very severe chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
A Multicentre, Parallel-group, Phase IIb, Randomised, Double-blind, Placebo-controlled, 4-Arm, 24-Week Study to Evaluate the Efficacy and Safety of AZD6793 Tablets in Adult Participants with Moderate to Very Severe Chronic Obstructive Pulmonary Disease (PRESTO)

Approximately 400 sites globally will participate in this study. Approximately 1160 participants will be randomized to four treatment groups; three different doses of AZD6793 vs placebo in a 1:1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥40 years of age at the time of signing the informed consent.
* Documented primary diagnosis of moderate to very severe COPD for at least 12 months prior to enrolment.
* Pre-BD FEV1/FVC < 0.7 at Visit 1 and pre- and post-BD FEV1/FVC < 0.7, and post-BD FEV1 ≥ 25% to < 80% of predicted normal at Visit 2.
* Documented history of ≥ 2 moderate or ≥ 1 severe COPD exacerbations in the 12 months prior to screening.
* Documented stable regimen of inhaled triple maintenance therapy or inhaled dual maintenance therapy for ≥ 3 months prior to screening.
* CAT score ≥ 10 at Visit 1.
* Current or ex-smokers with a cigarette smoking history of ≥ 10 pack-years.
* Participants who are clinically stable and free from an exacerbation of COPD for 4 weeks prior to Visit 1 and remain exacerbation free at Visit 3 (randomisation).
* Negative pregnancy test at Visit 1 and Visit 3 for Women Of Child-Bearing Potential (WOCBP).

Exclusion Criteria:

* Clinically important pulmonary disease other than COPD (eg, asthma [current diagnosis per GINA or other accepted guidelines], active pulmonary infection, clinically significant bronchiectasis when bronchiectasis is the predominant diagnosis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha-1 antitrypsin deficiency or primary ciliary dyskinesia).
* Radiological findings suggestive of a respiratory disease other than COPD that is significantly contributing to the participant's respiratory symptoms.
* Any unstable disorder, including, but not limited to, CV, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric disorder, major physical and/or cognitive impairment.
* Significant left heart failure.
* Unstable angina, acute coronary syndrome/acute myocardial infarction or coronary intervention with percutaneous coronary intervention/coronary artery bypass graft within 6 months of randomisation, uncontrolled arrhythmia, or cardiomyopathy, clinically significant aortic stenosis, or signs of pulmonary oedema or volume overload.
* Pulmonary arterial hypertension, either idiopathic or due to connective tissue or thromboembolic disease.
* History of another underlying condition that predisposes the participant to infections.
* History of ulcerative colitis, Crohn's disease, or microscopic colitis diagnosed by either a gastroenterologist or by histopathology.
* Abnormal laboratory findings.
* Participants with evidence of active liver disease and/or evidence of chronic liver disease.
* Participants with history of HIV infection or who test positive for HIV.
* History of lung volume reduction surgery.
* Current or history of malignancy within 5 years before the screening visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1160 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2027-11-05 (Estimated); Study Completion 2027-11-05 (Estimated)

PRIMARY OUTCOMES:
Annualised rate of moderate or severe COPD exacerbations | From baseline up to 24 Weeks
  The annualised moderate or severe COPD exacerbation rate (based on exacerbations reported by the investigator) up to 24 Weeks treatment period compared to placebo

SECONDARY OUTCOMES:
Time to first moderate or severe COPD exacerbation | From baseline up to 24 Weeks
  To evaluate the effect of AZD6793 as compared to placebo on COPD exacerbations from baseline up to 24 Weeks
Annualised rate of COPD exacerbations associated with emergency room visits, urgent care visits, or hospitalisations | From baseline up to 24 Weeks
  To evaluate the effect of AZD6793 as compared to placebo on COPD exacerbations from baseline up to 24 Weeks
Annualised rate of severe COPD exacerbations | From baseline up to 24 Weeks
  To evaluate the effect of AZD6793 as compared to placebo on COPD exacerbations from baseline up to 24 Weeks
Annualised rate of COPDCompEx events | From baseline up to 24 Weeks
  To evaluate the effect of AZD6793 as compared to placebo on COPDCompEx events from baseline up to 24 Weeks
Time to first COPDCompEx event | From baseline up to 24 Weeks
  To evaluate the effect of AZD6793 as compared to placebo on COPDCompEx events from baseline up to 24 Weeks
Change from baseline in pre-bronchodilator (pre-BD) forced expiratory volume in 1 second (FEV1) | From baseline to Week 12 and Week 24
  Change from baseline in pre-BD FEV1 at Week 12 and Week 24 compared to placebo
Change from baseline in post-bronchodilator (post-BD) forced expiratory volume in 1 second (FEV1) | From baseline to Week 12 and Week 24
  Change from baseline in post-BD FEV1 at Week 12 and Week 24 compared to placebo
Change from baseline in Breathlessness, Cough and Sputum Scale (BCSS) total score | From baseline over 24 Weeks
  Change from baseline in BCSS total score over 24 Weeks compared to placebo.
  The BCSS is a 3-item questionnaire rating breathlessness, sputum, and cough on a 5 point Likert scale from 0 (no symptoms) to 4 (severe symptoms). The BCSS has a scoring range of 0-12 with higher scores indicative of greater COPD impact on health status.
Change from baseline in COPD Assessment Test (CAT) total score | From baseline over 24 Weeks
  Change from baseline in the CAT total score over 24 weeks
  CAT is an 8-item PRO that measures the impact of COPD on the health status of patients with COPD. The CAT has a scoring range of 0-40 with higher scores indicative of greater COPD impact on health status.
Change from baseline in St George's Respiratory Questionnaire (SGRQ) total and domain scores | From baseline over 24 Weeks
  Participants achieving a clinically meaningful improvement from baseline in SGRQ total score (4-point score decrease) over 24 weeks.
  SGRQ is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with lower scores indicating better health status.
Measurement of plasma concentrations of AZD6793 at specific timepoints | From baseline to Week 4, Week 12 and Week 24
  To assess the pharmacokinetics (PK) of AZD6793 in participants with moderate to very severe COPD

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit, Manchester University NHS Foundations Trust, Manchester, United Kingdom
Locations (290):
- United States (73):
  - Research Site, Birmingham, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Canoga Park, California
  - Research Site, La Mesa, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Norco, California
  - Research Site, Tustin, California
  - Research Site, Lakewood, Colorado
  - Research Site, Brandon, Florida
  - Research Site, Cape Coral, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lake City, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Naples, Florida
  - Research Site, Ocala, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Plantation, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Suwanee, Georgia
  - Research Site, West Des Moines, Iowa
  - Research Site, Lexington, Kentucky
  - Research Site, Zachary, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Burlington, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Garden City, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Chesterfield, Missouri
  - Research Site, Hannibal, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Mount Kisco, New York
  - Research Site, New Bern, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, DuBois, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Scottdale, Pennsylvania
  - Research Site, Smithfield, Pennsylvania
  - Research Site, Lancaster, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Franklin, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, Denison, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Lewisville, Texas
  - Research Site, Mansfield, Texas
  - Research Site, McKinney, Texas
  - Research Site, Pearland, Texas
  - Research Site, Colchester, Vermont
  - Research Site, Norfolk, Virginia
  - Research Site, Williamsburg, Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Madison, Wisconsin
- Argentina (9):
  - Research Site, Alberdi
  - Research Site, CABA
  - Research Site, Capital Federal
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Ranelagh
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
- Australia (5):
  - Research Site, Cairns
  - Research Site, Norwood
  - Research Site, Osborne Park
  - Research Site, South Brisbane
  - Research Site, Wollongong
- Bulgaria (7):
  - Research Site, Dupnitsa
  - Research Site, Haskovo
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Veliko Tarnovo
  - Research Site, Yambol
- Canada (14):
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Truro, Nova Scotia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Stoney Creek, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Victoriaville, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Chile (6):
  - Research Site, Chile
  - Research Site, Concepción
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (22):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hohhot
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Wuhan
  - Research Site, Xuzhou
  - Research Site, Zhengzhou
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Esbjerg
  - Research Site, Hvidovre
  - Research Site, Odense C
  - Research Site, Roskilde
- Germany (15):
  - Research Site, Ahrensburg
  - Research Site, Bendorf
  - Research Site, Berlin
  - Research Site, Darmstadt
  - Research Site, Halle
  - Research Site, Hanover
  - Research Site, Landsberg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Marburg
  - Research Site, Obertshausen
  - Research Site, Rosenheim
  - Research Site, Schleswig
  - Research Site, Wiesbaden
  - Research Site, Witten
- Greece (3):
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Thessaloniki
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Edelény
  - Research Site, Encs
  - Research Site, Gödöllő
  - Research Site, Hajdúnánás
  - Research Site, Nyíregyháza-Sóstóhegy
  - Research Site, Törökbálint
- India (9):
  - Research Site, Belagavi
  - Research Site, Coimbatore
  - Research Site, Dehradun
  - Research Site, Dwārka
  - Research Site, Hyderabad
  - Research Site, Kochi
  - Research Site, Mumbai
  - Research Site, Nagpur
  - Research Site, Vijayawada
- Italy (9):
  - Research Site, Busto Arsizio
  - Research Site, Cuneo
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Statte
  - Research Site, Telese Terme
- Japan (35):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Ginowan-shi
  - Research Site, Hachioji-shi
  - Research Site, Hamamatsu
  - Research Site, Hiroshima
  - Research Site, Izumi-shi
  - Research Site, Kamakura
  - Research Site, Kanazawa
  - Research Site, Kasuga-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kiyosu-shi
  - Research Site, Kochi
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Matsuyama
  - Research Site, Minoh
  - Research Site, Minokamo Shi
  - Research Site, Mizunami-shi
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Sasebo-shi
  - Research Site, Shimotsuga-gun
  - Research Site, Shinjuku-ku
  - Research Site, Tachikawa-shi
  - Research Site, Toon-shi
  - Research Site, Toyota
  - Research Site, Ube
  - Research Site, Yokkaichi-shi
  - Research Site, Yokohama
- Mexico (5):
  - Research Site, Chihuahua City
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Monterrey
- Research Site, Lima, Peru
- Poland (16):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Chęciny
  - Research Site, Elblag
  - Research Site, Karczew
  - Research Site, Katowice
  - Research Site, Komorniki
  - Research Site, Ksawerów
  - Research Site, Lodz
  - Research Site, Ostróda
  - Research Site, Piaseczno
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Warsaw
- South Korea (8):
  - Research Site, Anyang-si
  - Research Site, Cheongju-si
  - Research Site, Chuncheon
  - Research Site, Daegu
  - Research Site, Jeonju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Wŏnju
- Spain (7):
  - Research Site, Benalmádena
  - Research Site, Granollers
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Mérida
  - Research Site, Pozuelo de Alarcón
  - Research Site, Santander
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yung Kang City
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, İzmit
  - Research Site, Kayseri
  - Research Site, Mersin
- Ukraine (6):
  - Research Site, Chernivtsi
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Ternopil
  - Research Site, Uzhhorod
- United Kingdom (8):
  - Research Site, Bradford
  - Research Site, Cottingham
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Thetford
  - Research Site, Wythenshawe
- Vietnam (6):
  - Research Site, Da Nang
  - Research Site, Dong Thập
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Huế
  - Research Site, Rach Gia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/